CLINICAL TRIAL: NCT03066518
Title: A Randomized Placebo-controlled Trial Evaluating the Effect of Melatonin on Sleep Quality in Patients With Dementia
Brief Title: Effect of Melatonin on Sleep Quality in Patients Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Rocio Morales Delgado, MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE15-002
Record Dates: First submitted 2017-02-19; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Sleep Disorders; Dementia
Keywords: melatonin; sleep; dementia; cognition
MeSH Terms: conditions — Sleep Wake Disorders; Dementia | interventions — Melatonin; pyrithyldione

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Selection for a treatment group was determined by a computer-generated randomization list, in a 1:1 ratio using the randomized permuted blocks method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Placebo Comparator): Melatonin 5 mg, daily, eight weeks
  Interventions: Drug: Melatonin 5 mg
- placebo (Placebo Comparator): Placebo, daily, eight weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin 5 mg
  Other Names: Benedorm
  Arms: Melatonin
Other: Placebo
  Arms: placebo

SUMMARY:
Introduction: Patients with dementia may suffer from poor sleep quality. Disturbance in the metabolism melatonin may have a role in the pathogenesis of sleep-wake cycle alterations in dementia.

Objective: To evaluate the efficacy of low dose exogenous melatonin in improving sleep quality.

Design: A single-center randomized, double-blinded, placebo-controlled study carried out on outpatients with dementia and sleep alterations.

Participants: The investigators calculated a 40 individuals aged 65 years or over with a diagnosis of mild-moderate dementia (Clinical Dementia Rating 1-2).

Intervention: Patients were randomized to receive either 5 mg of melatonin or placebo every night for 8 weeks.

Measurements: The primary outcome was sleep quality according to the Pittsburgh Sleep Quality Index (PSQI).

DETAILED DESCRIPTION:
This is a single-center study. The study protocol, informed consents, and amendments were approved in writing by the appropriate local site Independent Ethics Committee (IEC)/Institutional Review Boards (IRB) (Ethics Committee of the Universidad Autónoma de Nuevo León, School of Medicine).

The patients were recruited as outpatients from the Geriatrics Clinic. A total of 67 patients were screened out of which 40 male and female patients diagnosed with mild to moderate dementia were recruited to the study. Following inclusion, all patients underwent randomization to treatment with melatonin (5 mg orally) or placebo for 8 weeks. To prevent bias, matching placebo tablets, which were identical in appearance, taste, and odor, were used. The treatment was double-blinded, with two parallel treatment groups. Selection for a treatment group was determined by a computer-generated randomization list, in a 1:1 ratio using the randomized permuted blocks method.

ELIGIBILITY:
Inclusion Criteria:

* Older than 60 years;
* Circadian cycle sleep disorder with insomnia (according to Diagnostic and Statistical Manual of Mental Disorders- V criteria);
* Mild or moderate dementia (clinical dementia rating 1 and 2);
* Medications such as anti-depressants, acetylcholinesterase inhibitors, antipsychotics or memantine were allowed as long as they were initiated for over 8 weeks.

Exclusion Criteria:

* They had other diagnoses of sleep disorders, known hypersensitivity to melatonin, use of stimulants or hypnotics, recent diagnosis (within 8 weeks) of mood disorders or neuropsychiatric symptoms.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 8 weeks
  A self-administered questionnaire that provides an overall rating of sleep quality.

SECONDARY OUTCOMES:
Minimental test | baseline and to the 8 weeks
  The original purpose is to allow physicians to standardize and quantify cognitive status.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Guajardo, MD, Study Director — HUGonzález

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Crowley K. Sleep and sleep disorders in older adults. Neuropsychol Rev. 2011 Mar;21(1):41-53. doi: 10.1007/s11065-010-9154-6. Epub 2011 Jan 12. PMID 21225347
- [Background] Neikrug AB, Ancoli-Israel S. Sleep disorders in the older adult - a mini-review. Gerontology. 2010;56(2):181-9. doi: 10.1159/000236900. Epub 2009 Sep 9. PMID 19738366
- [Background] Beaulieu-Bonneau S, Hudon C. Sleep disturbances in older adults with mild cognitive impairment. Int Psychogeriatr. 2009 Aug;21(4):654-66. doi: 10.1017/S1041610209009120. Epub 2009 May 11. PMID 19426575
- [Background] Woods DL, Phillips LR, Martin JL. Biological basis for sleep disturbance and behavioral symptoms in dementia: a biobehavioral model. Res Gerontol Nurs. 2011 Oct;4(4):281-93. doi: 10.3928/19404921-20110302-01. Epub 2011 Mar 16. PMID 21417189
- [Background] Guarnieri B, Cerroni G, Sorbi S. Sleep disturbances and cognitive decline: recommendations on clinical assessment and the management. Arch Ital Biol. 2015 Jun-Sep;153(2-3):225-30. doi: 10.12871/0003982920152347. PMID 26742676
- [Background] Ooms S, Ju YE. Treatment of Sleep Disorders in Dementia. Curr Treat Options Neurol. 2016 Sep;18(9):40. doi: 10.1007/s11940-016-0424-3. PMID 27476067
- [Background] Xu J, Wang LL, Dammer EB, Li CB, Xu G, Chen SD, Wang G. Melatonin for sleep disorders and cognition in dementia: a meta-analysis of randomized controlled trials. Am J Alzheimers Dis Other Demen. 2015 Aug;30(5):439-47. doi: 10.1177/1533317514568005. PMID 25614508
- [Background] McCleery J, Cohen DA, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2016 Nov 16;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub3. PMID 27851868
- [Background] Chien MY, Chen HC. Poor sleep quality is independently associated with physical disability in older adults. J Clin Sleep Med. 2015 Mar 15;11(3):225-32. doi: 10.5664/jcsm.4532. PMID 25515275
- [Derived] Morales-Delgado R, Camara-Lemarroy CR, Salinas-Martinez R, Gamez-Trevino D, Arredondo-Jaime A, Hernandez-Maldonado E, Guajardo-Alvarez G. A randomized placebo-controlled trial evaluating the effect of melatonin on sleep quality in patients with mild-moderate dementia. Eur Geriatr Med. 2018 Aug;9(4):449-454. doi: 10.1007/s41999-018-0068-9. Epub 2018 May 24. PMID 34674490
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083